CLINICAL TRIAL: NCT04134208
Title: 18F-Fluciclovine PET CT as an Indicator of Therapeutic Response in Metastatic Prostate Carcinoma (M1PCa)
Brief Title: An Investigational Scan (18F-Fluciclovine PET-CT) for the Measurement of Therapeutic Response in Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0030; NCI-2019-06047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0030 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fluciclovine F18, PET-CT) (Experimental): Within 4 weeks before starting SST, patients receive fluciclovine F18 IV then undergo a PET-CT scan over 30 minutes. Within 22-28 weeks after starting SST, patients receive fluciclovine F18 IV and undergo a second PET-CT scan over 30 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Fluciclovine F18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET-CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Procedure: Positron Emission Tomography — Undergo PET-CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase IV trial studies how well an investigational scan (18F-fluciclovine PET-CT) works for the measurement of therapeutic response in patients with prostate cancer that has spread to other places in the body (metastatic). 18F-fluciclovine is a radioactive substance that is used in this study with PET-CT imaging scans that may help doctors learn about response to standard therapy in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate metabolic response by fluciclovine F18 (18F-fluciclovine) PET qualitatively and semi-quantitatively with standardized uptake values (SUV) following androgen deprivation therapy (ADT) plus abiraterone at 22-28 weeks (+/- 4 weeks), and correlate the findings with size changes as defined by conventional imaging and prostate-specific antigen (PSA) response.

SECONDARY OBJECTIVES:

I. To correlate pelvic 18F-fluciclovine PET imaging findings with pathologic findings at radical prostatectomy and pelvic lymph node dissection to determine 18F-fluciclovine PET imaging sensitivity and specificity for pelvic lymph node cancer involvement.

II. To evaluate 18F-fluciclovine PET imaging response and its correlation with progression free survival (defined by Prostate Cancer Working Group 2 [PCWG2] criteria).

III. To determine if sites of progressive disease develop at the initial/prior site (diagnostic site) of metastases or in newly developed sites at the time of metastatic progression.

IV. To evaluate metabolic response by 18F-fluciclovine PET semi-quantitatively with target to blood pool ratio (TBR) following ADT plus abiraterone at 22-28 weeks (+/- 4 weeks), and correlate the findings with size changes as defined by conventional imaging and PSA response.

OUTLINE:

Within 4 weeks before starting standard systemic therapy (SST), patients receive fluciclovine F18 intravenously (IV) then undergo a PET-CT scan over 30 minutes. Within 22-28 weeks after starting SST, patients receive fluciclovine F18 IV and undergo a second PET-CT scan over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven prostate carcinoma
* Documented evidence of M1 disease by American Joint Committee on Cancer (AJCC) staging by bone scan, CT and magnetic resonance imaging (MRI)
* Castration naive disease, no prior systemic therapy for prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to understand and willingness to sign informed consent

Exclusion Criteria:

* Known brain metastasis
* Small cell carcinoma of the prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Ravizzini, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical Clinic
Pre-assignment Details: No enrolled participants were excluded from the study
Period: Overall Study
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Median (Standard Deviation); unit: years] | 70.5 (70.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Response by Fluciclovine F18 (18F-fluciclovine) Positron Emission Tomography (PET) With Standardized Uptake Values (SUV)"
Description: Will evaluate metabolic response by 18F-fluciclovine PET qualitatively and semi-quantitatively with SUV and correlate the findings with size changes as defined by conventional imaging prostate specific antigen (PSA) response. The percentage of change in the 18F-fluciclovine maximum standardized uptake value (SUVmax) after therapy will be calculated as follows ([pretreatment corrected SUVmax - posttreatment corrected SUVmax]/pretreatment corrected SUVmax) x 100. Similar calculations will be performed for mean SUV, metabolic tumor volume, and total volume activity.
  An analysis of the quantitative data was recently performed for the 2 participants.
Time Frame: Up to 2 years
Population: No ROC analysis was performed due to the small number of patients. An analysis of the quantitative data was recently performed.
Measure: Number; unit: percentage of change
Groups:
- Diagnostic (Fluciclovine F18, PET-CT) (Participant #1); Diagnostic (Fluciclovine F18, PET-CT) (Participant #2): Within 4 weeks before starting SST, patients receive fluciclovine F18 IV then undergo a PET-CT scan over 30 minutes. Within 22-28 weeks after starting SST, patients receive fluciclovine F18 IV and undergo a second PET-CT scan over 30 minutes.
  Computed Tomography: Undergo PET-CT scan
  Fluciclovine F18: Given IV
  Positron Emission Tomography: Undergo PET-CT scan
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT) (Participant #1) | Diagnostic (Fluciclovine F18, PET-CT) (Participant #2)
Number analyzed (Participants) | 1 | 1
percentage of change
  SUVmax | -69.9 | -50
  SUVmean | -46.3 | -37.5

2. Secondary Outcome: 18F-fluciclovine PET Imaging Response - SUVMax
Description: Will evaluate 18F-fluciclovine PET imaging response and its correlation with progression free survival defined by Prostate Cancer Working Group 2 criteria.
Time Frame: Up to 2 years
Population: We compare F-18 fluciclovine PET/CT uptake (SUVmax) in tumors before and after treatment.
Measure: Number; unit: ng/mL
Groups:
- Diagnostic (Fluciclovine F18, PET-CT) Participant #1; Diagnostic (Fluciclovine F18, PET-CT) Participant #2: Within 4 weeks before starting SST, patients receive fluciclovine F18 IV then undergo a PET-CT scan over 30 minutes. Within 22-28 weeks after starting SST, patients receive fluciclovine F18 IV and undergo a second PET-CT scan over 30 minutes.
  Computed Tomography: Undergo PET-CT scan
  Fluciclovine F18: Given IV
  Positron Emission Tomography: Undergo PET-CT scan
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT) Participant #1 | Diagnostic (Fluciclovine F18, PET-CT) Participant #2
Number analyzed (Participants) | 1 | 1
ng/mL
  SUVmax baseline | 10.8 | 6.6
  SUVmax posttreatment | 4.1 | 3.3

3. Secondary Outcome: 18F-fluciclovine PET Imaging Response - SUVMean
Description: Will evaluate 18F-fluciclovine PET imaging response and its correlation with progression free survival defined by Prostate Cancer Working Group 2 criteria. SUVmean represents the average SUV value across a defined region of interest (ROI) in the tumor. The Measure Type is a number, that is dimensionless, because it is the average ratio of tissue activity concentration to the injected dose normalized by the patient's weight.
Time Frame: Up to 2 years
Population: We compare F-18 fluciclovine PET/CT uptake (SUVmean) in tumors before and after treatment.
Measure: Number; unit: mg/mL
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT) Participant #1 | Diagnostic (Fluciclovine F18, PET-CT) Participant #2
Number analyzed (Participants) | 1 | 1
mg/mL
  SUVmean baseline | 4.9 | 5.2
  SUVmean posttreatment | 3.2 | 3.3

4. Secondary Outcome: 18F-fluciclovine PET Imaging Response - Metabolic Tumor Volume
Description: as for outcome 2
Time Frame: Up to 2 years
Population: We compare F-18 fluciclovine PET/CT uptake (Metabolic Tumor Volume) in tumors before and after treatment.
Measure: Number; unit: mL
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT) Participant #1 | Diagnostic (Fluciclovine F18, PET-CT) Participant #2
Number analyzed (Participants) | 1 | 1
mL
  metabolic tumor volume baseline | 33.6 | 1.2
  metabolic tumor volume posttreatment | 0.5 | 0.03

5. Secondary Outcome: Sites of Progressive Disease Development
Description: Will determine if sites of progressive disease develop at the initial/prior site (diagnostic site) of metastases or in newly developed sites at the time of metastatic progression.
Time Frame: Up to 2 years
Population: No newly developed sites of disease were identified (no progressive disease). The primary prostate tumors were biopsied pretreatment, but not re-biopsied post-treatment. In patient#1, a left common iliac lymph node was biopsied prior to treatment, but not re-biopsied after treatment, since this lymph node resolved posttreatment. No analysis for sensitivity and specificity were performed.
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT)
Number analyzed (Participants) | 0

6. Secondary Outcome: Metabolic Response by 18F-fluciclovine PET With Target to Blood Pool Ratio (TBR)
Description: Will evaluate metabolic response by 18F-fluciclovine PET semi-quantitatively with TBR and correlate the findings with size changes as defined by conventional imaging and PSA response.
Time Frame: Up to 2 years
Population: Participant #1 underwent baseline imaging, first post-treatment and second post-treatment PET CT scans. Participant #1 second post-treatment data were not measured, since there was no "target." There was no site of disease present on the second posttreatment scan, lesions resolved.
  The #2 patient did not have any second posttreatment scan.
Measure: Number; unit: target to blood ratio (TBR)
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT) (Participant #1) | Diagnostic (Fluciclovine F18, PET-CT) (Participant #2)
Number analyzed (Participants) | 1 | 1
target to blood ratio (TBR)
  Baseline | 7.66 | 4.85
  First post-treatment | 1.19 | 2.04
  Second post-treatment: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Description: No Adverse Events were observed or reported
Arm/Group | Diagnostic (Fluciclovine F18, PET-CT)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT04134208/Prot_SAP_006.pdf
  • Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT04134208/ICF_007.pdf